CLINICAL TRIAL: NCT02664844
Title: Physical Activity and Food Intake Interaction: Effect of Weight Loss in Obese Adolescent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0255
Record Dates: First submitted 2016-01-15; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: Obesity; Appetite regulation; Insulin sensitivity; Adolescents; Exercise
MeSH Terms: conditions — Obesity; Insulin Resistance; Motor Activity | interventions — Exercise

ARMS (1):
- Obese adolescent (Experimental)
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity

SUMMARY:
In obese adolescents, energy expenditure (EE) of chronic high intensity muscular exercise (> 70% VO2max) conducted one hour before a meal causes an anorectic effect at lunch and dinner the same day. The effect on food intake of the distribution of this exercise into two sessions during 24h remains to be determined. In addition, a multidisciplinary load of obesity generates a loss of body weight in the short term, which we do not know the effects on energy balance. To our knowledge, the impact of weight loss on the anorectic effect of muscle exercise is unknown.

DETAILED DESCRIPTION:
Two measuring sequences will be carried out before (M0) and after 4 months (M4) of a multidisciplinary treatment program of four months. Each sequence will have three days: a "sedentary" day (SED) and two days "exercise" (EX). During the exercise day "EX1", a continuous intense exercise will be conducted for 40 min at 70% VO2max of subjects. During the second day exercise "EX2" teenage realize two exercise representing the same DE as EX1 in the morning (50% ED) and late afternoon (50% ED). The multidisciplinary management program (without energy restriction) controlled by institution consists of nutrition education, physical activity and therapeutic education. The exercise program will involve the activity sessions controlled and supervised by a sports educator and interactive sessions using a scientifically validated physical activity program (Biomouv®).

ELIGIBILITY:
Inclusion Criteria:

* Overweight adolescents (over the 90 th percentile of the international cut-off point)
* Sedentary (according to the IPAQ-A questionnaire)
* Without eating disorders (according to the DEBQ questionnaire)

Exclusion Criteria:

* Medical or surgical antecedents that are incompatible with the study: cardiovascular, endocrine or digestive disease.
* Drugs that could interfere with the results of the study
* Surgical intervention in the 3 months
* Regular consumption of tobacco or Alcohol
* patients on a diet with caloric restriction
* Refusal to sign the consent form
* Regular practice of sport and intensive

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Comparison between(M0) and (M4) of food intake on 24 hours (total and per meal) | after 4 months of physical activity
  Comparison between(M0) and (M4) of food intake on 24 hours (total and per meal) assessed during a day with the completion of intense exercise performed in one session EX1, in two sessions (EX2) or sedentary (without exercise: SED). The exercise-induced energy expenditure by 40 minutes at 70% of VO2 max is the same in EX1 and EX2.

SECONDARY OUTCOMES:
Comparison between(M0) and (M4) of the Flint scale | after 4 months of physical activity
  Comparison between(M0) and (M4) of the Flint scale (feeling of hunger, desire to eat, the feeling of being full)
Comparison between(M0) and (M4) of the Pittsburg scale | after 4 months of physical activity
Comparison between(M0) and (M4) of HOMA-IR | after 4 months of physical activity
  Comparison between(M0) and (M4) of HOMA-IR by measuring the blood glucose and fasting insulin
Comparison between(M0) and (M4) of Fitness | after 4 months of physical activity
  Comparison between(M0) and (M4) of Fitness (by VO2 max and estimated body composition).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France